CLINICAL TRIAL: NCT05881850
Title: The Effect of the Education Program on Increasing Osteoporosis Awareness Given to Women Aged 18-49 on Osteoporosis Awareness and Osteoporosis Health Beliefs
Brief Title: Education Program on Increasing Osteoporosis Awareness Given to Women Aged 18-49
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Melike Erguven Boga, Registered nurse, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 861123-11/658
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis Risk
Keywords: Osteoporosis; Osteoporosis Health Belief; Awareness; Education Program; Women Health
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The research will be conducted in a pre-test-post-test order, as a randomized controlled experimental.
Who Masked: Outcomes Assessor
Masking Description: The statistical expert who performs the randomization of the study and the statistical expert who evaluates the pre- and post-intervention data obtained in the study are different from each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): After the participants are given the necessary information about the research and written consent is obtained, the introductory information form, Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied by the researcher to the women in the intervention group who meet the inclusion criteria in the study to collect pre-test data just before the education program begins. Twelve weeks after finishing the education program the Osteoporosis Awareness Scale and the Osteoporosis Health Belief Scale will be administered to collect the posttest data.
  Interventions: Other: Education Program on Increasing Osteoporosis Awareness Given to Women Aged 18-49. The research is carry out as a randomized controlled experimental in a pretest-posttest design.
- Control group (No Intervention): After the participants were given the necessary information about the study and written consents were obtained, the Introductory Information Form, Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied to the women in the control group who met the inclusion criteria in order to collect the pre-test data. Twelve weeks after finishing the education program, the Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied to collect the post-test data.

INTERVENTIONS:
Other: Education Program on Increasing Osteoporosis Awareness Given to Women Aged 18-49. The research is carry out as a randomized controlled experimental in a pretest-posttest design. — The education program consisting of three sessions was held once a week and each session lasted approximately 40-50 minutes. In the realization of the education program, a power point presentation consisting of the contents of the education booklet prepared for Osteoporosis awareness, a three-dimensional bone model with Osteoporosis and normal bone tissue, some food samples containing calcium during nutrition education, and measuring cups to show portions and amounts were used. During the training, a question and answer activity was also held. The education booklet was also given to the intervention group at the end of the first session.
  Arms: Intervention group

SUMMARY:
Summary Purpose: To examine the effect of the education program to increase osteoporosis awareness given to women aged 18-49.

The research is carry out as a randomized controlled experimental in a pretest-posttest design. The population of the research consisted of women registered in four different women's cultural and education centers affiliated with Ankara Altındağ Municipality between the dates of data collection.The number of women to be included in the sample of the study was determined as 70 women, 35 of which were in the control group, in the analysis made using the G*Power 3.1.9.2 program. Intervention and control groups were assigned to the groups by randomization method. The data collection tools used in the research are the Introductory Information Form, the Osteoporosis Health Belief Scale and the Osteoporosis Awareness Scale. In the implementation of the research, the education program to increase awareness of osteoporosis was carried out on certain days of the week with groups of at least two and at most five women. The education program aimed at raising awareness of osteoporosis was carried out in 3 sessions, one week apart, and each session lasted approximately 40-50 minutes. Before the first session of the education program, pre-test data were collected from the intervention and control groups. Post-test data will be collected through the Osteoporosis Health Belief Scale and the Osteoporosis Awareness Scale from women in the intervention and control groups twelve weeks after finishing the education program.

DETAILED DESCRIPTION:
Type of Research The research will be conducted as a randomized controlled experimental study in the pre-test-post-test order.

Research hypotheses H11 : There is a difference between the osteoporosis awareness scores of the women who participated in the training program to increase the awareness of osteoporosis and the osteoporosis awareness scores of the women who did not participate in the training program.

H01: There is no difference between the osteoporosis awareness scores of the women who participated in the training program to increase the awareness of osteoporosis and the osteoporosis awareness scores of the women who did not participate in the training program.

H12: There is a difference between the osteoporosis health belief scores of women who participated in the training program to increase awareness of osteoporosis and the osteoporosis health belief scores of women who did not participate in the training program.

H02: There is no difference between the osteoporosis health belief scores of the women who participated in the training program to raise awareness of osteoporosis and the osteoporosis health belief scores of the women who did not attend the training.

Place of Research

The research is planned to be carried out in the Women's Culture and Education Centers of Ankara Altındağ Municipality. Altındağ Municipality has 24 Women's Culture and Education Centers in 24 different neighborhoods with a total of 60000 registered members (https://www.altindag.bel.tr/#!kadin_egitim_kultur_merkezleri). The research was conducted in the first four centers with the highest number of members among the 24 Women's Culture and Education Centers. Necessary permissions were obtained from the centers where the research would be conducted. The permission obtained was reported to the Ethics Committee.

Population and Sample of the Research

In this study, the G*Power-3.1.9.2 program was used to calculate the sample size. The sample size was calculated at a 95% confidence level based on the Osteoporosis Health Belief Scale scores as a result of the study conducted by Pınar and Pınar (2020). As a result of the analysis, α=0.05 level, standardized effect size was calculated as d=0.9530, and with a power of 0.95, a minimum of 60 women, 30 in the intervention group and 30 in the control group, were found.

Considering the possibility of participants who did not want to continue with the research, the number of women to be included in the sample of the study was determined as 70, taking into account the dropout rate of a similar study (Eyimaya & Tezel, 2021). According to the results of the power analysis, intervention and control groups will be determined by randomization among women who meet the inclusion criteria and agree to participate in the study.

The managers of the institutions in the centers where the research will be conducted made an announcement about osteoporosis awareness training to women aged between 18-49, and the women were invited to the research and a list of volunteers was created. The researcher contacted the volunteer women and identified the women who met the inclusion criteria in the study. The list of the volunteers who met the criteria for inclusion in the study, including their age, educational status and the center they were a member of, was sent to a statistics expert in order to determine the intervention and control groups by randomization method.

Data Collection Tools Introductory Information Form Osteoporosis Awareness Scale Osteoporosis Health Belief Scale

Introductory Information Form

In order to determine the introductory characteristics of the participants (age, educational status, etc.), a form was prepared by the researcher using the literature. The form was presented to the opinion of 6 different experts who are faculty members in the fields of Gynecology and Obstetrics Nursing, Midwifery, Nutrition and Dietetics, Physiotherapy and Rehabilitation and was arranged according to their suggestions.

Osteoporosis Awareness Scale

The Osteoporosis Awareness Scale was developed by Choi et al. (2008). In the original version of the scale, there are 31 questions and sub-dimensions of "protective behaviors", "risk factors", "characteristics of osteoporosis", "bone physiology" and "improving bone health". Turkish validity and reliability studies of the scale were performed by Aktürk et al. (2021). In the Turkish version of the scale, the "improving bone health" sub-dimension in the original scale was not included, but the "exercise" sub-dimension was included. However, the number of questions has been reduced to 27. The sub-dimensions in the Turkish form of the scale are; "protective behaviors", "risk factors", "characteristics of osteoporosis", "exercise" and "bone physiology".

Cronbach's alpha value of the scale was 0.948 and sub-dimension Cronbach's alpha values; 0.917 for "protective behaviors", 0.820 for "risk factors", 0.839 for "osteoporosis features", 0.821 for "bone physiology" and 0.804 for "bone health promotion". In the adaptation study of the scale to Turkish society, Cronbach's alpha value was 0.949 and sub-dimension Cronbach's alpha values; It was found to be 0.86 for "protective behaviors", 0.866 for "bone physiology", 0.882 for "risk factors", 0.866 for "exercise" and 0.858 for "characteristics of osteoporosis".

Osteoporosis Health Belief Scale

The Osteoporosis Health Belief Scale was developed by Kim et al. (1991) to measure health beliefs about osteoporosis based on the Health Belief Model. The Turkish validity and reliability analyzes of the scale were performed by Kılıç and Erci (2004). There are 42 questions and seven sub-dimensions in the scale. The sub-dimensions of the scale are "perception of sensitivity", "perception of seriousness", "benefits of exercise", "benefits of taking calcium", "barriers to exercise", "obstacles of calcium intake" and "health motivation". The Cronbach's alpha value of the scale is between 0.71-0.82 (Kim et al., 1991). The Cronbach alpha value of the scale, which was adapted into Turkish, is between 0.79-0.94.

Education Program to Raise Osteoporosis Awareness

The education program was prepared using the relevant literature, and the content of the training program was presented to the opinion of experts in the field and arranged according to their suggestions. Before starting the research, a preliminary application of the education program was carried out with three volunteer women who were randomly selected from the universe and met the criteria for inclusion in the sampling in a women's cultural center affiliated with Altındağ Municipality and for which data was not collected.

The education program, which was prepared to increase awareness of osteoporosis, was planned to be one-to-one education for each woman instead of group training due to the pandemic conditions, but on 05.05.2023 the World Health Organization and T.R. Following the Ministry of Health's notification that the Covid-19 global emergency has ended and the request from the participants in the pre-implementation of the education program, an application was made to the Ankara University Ethics Committee, and the necessary permission was obtained for the education to be implemented as a group training instead of one-on-one. However, permission was obtained from the Ethics Committee to reduce the time between education sessions to one week without changing the number of sessions.

The education program consisting of three sessions was held once a week and each session lasted approximately 40-50 minutes. In the realization of the education program, a power point presentation consisting of the contents of the education booklet prepared for Osteoporosis awareness, a three-dimensional bone model with Osteoporosis and normal bone tissue, some food samples containing calcium during nutrition education, and measuring cups to show portions and amounts were used. During the training, a question and answer activity was also held. The education booklet was also given to the intervention group at the end of the first session.

Contents of the Education Booklet

A education booklet will be used in the education to be given during the implementation of the education program to increase awareness of osteoporosis. The education booklet was created in line with the relevant literature. It was sent to a total of 6 experts who are faculty members of the field of Gynecology and Obstetrics Nursing, Midwifery, Nutrition and Dietetics, Physiotherapy and Rehabilitation for evaluation. The education booklet presented to the expert opinions was also evaluated according to the DISCERN measurement tool. In our study, after the evaluation of the education booklet, the DISCERN score average was calculated as 72.5. The readability coefficient of the education booklet was calculated according to Ateşman's (1997) formula. According to the calculations made, the readability coefficient of the education Manual for Raising Osteoporosis Awareness for Women aged 18-49 was calculated as 67.7. It indicates that the readability level of this booklet is medium difficulty.

Data Collection

Collection of intervention group data

After giving the necessary information about the research to the participants and obtaining written permissions, an introductory information form, Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied by the researcher to the women in the intervention group who meet the inclusion criteria, just before the education program (before first session) in order to collect the pre-test data. Six weeks after the pre-test data were collected, the Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied to collect the post-test data. In the awareness studies in the literature, studies measuring post-test data 15 days after the intervention or at wider time intervals were found (Alnuaimi et al., 2021; Erenoğlu and Yaman Sözbir, 2020; Darawad et al., 2022). In this study, a study measuring twelve weeks later was taken as reference (Öz Yıldırım et al., 2023).

Collection of control group data

After the participants were given the necessary information about the study and written consents were obtained, the Introductory Information Form, Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied to the women in the control group who met the inclusion criteria in order to collect the pre-test data.Twelve weeks after finishing the education program the Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale will be applied to collect the post-test data.

Variables of the Study

Dependent variable: Osteoporosis awareness and Osteoporosis health belief. Independent variable: Education program to raise awareness of osteoporosis.

Analysis of Data SPSS (Statistical Package for Social Sciences) program will be used to evaluate the data obtained from the research. In the analysis of continuous variables obtained from the measurements, mean and standard deviation, median (min-max), frequency and percentage values will be used in the analysis of categorical variables. It will be evaluated whether the continuous variables comply with the normal distribution by analyzing whether they comply with the parametric test conditions.

The average score will be taken in the evaluation of the scales. In order to compare the research groups, Student's t test will be used in cases where normal distribution is provided, and Mann-Whitney U test will be used in cases where normal distribution is not provided. In the analysis of the difference between the pre-test and post-test scores of the participants, appropriate tests will be performed after determining whether the data are suitable for normal distribution. Cronbach's alpha reliability coefficient will be calculated in the internal consistency analyzes of the scales and the reliability of their sub-dimensions. In all statistical analyzes, p values less than 0.05 will be considered statistically significant.

Ethical Principles Permission was obtained from the Ankara University Ethics Committee to conduct the study. The necessary permissions from the centers where the research will be conducted were obtained within the scope of the cooperation protocol between Ankara University Nursing Faculty and Altındağ Municipality. The permission obtained was reported to the Ethics Committee. In order to use the scales to be used in the research, permission was obtained from the authors via e-mail. Participants included in the study will be informed about the research through the Informed Voluntary Consent Form, and will be included in the study after their written consents are obtained.

After the education program given to the women in the intervention group is over, the women in the control group and all the women who volunteered to participate in the research but were not in the control or intervention groups will be given a education and a education booklet, consisting of one session, in three groups.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-49,
* Volunteering to participate in the study,
* To be at least primary school graduate,
* Not being pregnant or breastfeeding
* Not having a condition that prevents him from exercising,
* Not having a diet that limits daily calcium needs,
* Not having a planned training on osteoporosis before,
* Not being diagnosed with osteoporosis or osteopenia,
* Not be in the menopausal period,
* Not having a chronic disease
* Not having a situation that prevents communication (vision, hearing impairment, etc.).

Exclusion Criteria:

* Not participating in the entire training program,
* Failure to fill in all of the data collection tools during the research process.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Pre-test data: An introductory information form, Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale | just before the education program (before first session)
  1. Osteoporosis Awareness Scale: There are 27 questions and five sub-dimensions in the scale. The items in the scale are in four-point Likert type and classified as "I don't know at all" = 1, "I know a little" = 2, "I know" = 3, "I know very well" = 4. There are no reverse items and cut-off points in the scale. The total score obtained from the scale is minimum=27 maximum=108. As the score obtained from the scale increases, the level of awareness towards osteoporosis increases (Aktürk et al., 2021).
  2. There are 42 questions and seven sub-dimensions in the scale. The items in the scale are five-point Likert type, and the answer "strongly disagree"=1, "disagree" =2, "undecided" =3, "agree"=4, and "strongly agree" is evaluated as 5 points.The lowest score that can be obtained from the scale is 42 and the highest score is 210. The high score of the scale directly affects the health protective and improving behaviors of the person (Kılıç and Erci, 2004).

SECONDARY OUTCOMES:
Post-test data: Osteoporosis Awareness Scale and Osteoporosis Health Belief Scale | Eight weeks after the pre-test data were collected
  1. Osteoporosis Awareness Scale: There are 27 questions and five sub-dimensions in the scale. The items in the scale are in four-point Likert type and classified as "I don't know at all" = 1, "I know a little" = 2, "I know" = 3, "I know very well" = 4. There are no reverse items and cut-off points in the scale. The total score obtained from the scale is minimum=27 maximum=108. As the score obtained from the scale increases, the level of awareness towards osteoporosis increases (Aktürk et al., 2021).
  2. There are 42 questions and seven sub-dimensions in the scale. The items in the scale are five-point Likert type, and the answer "strongly disagree"=1, "disagree" =2, "undecided" =3, "agree"=4, and "strongly agree" is evaluated as 5 points.The lowest score that can be obtained from the scale is 42 and the highest score is 210. The high score of the scale directly affects the health protective and improving behaviors of the person (Kılıç and Erci, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Funda Ozturk, Assos. Prof., Study Director — Ankara University
Locations (1):
- Altındağ Municipality; Karapürçek 1, Mimar Başak Cengiz, Yıldıztepe, Beşikkaya Women's Culture and Education Centers, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eyimaya AO, Tezel A. The effect of nursing approaches applied according to Meleis' Transition Theory on menopause-specific quality of life. Health Care Women Int. 2021 Jan;42(1):107-126. doi: 10.1080/07399332.2020.1825440. PMID 33764278
- [Result] Choi E, Kim J, Chung M, Hwang K. [Development of an osteoporosis awareness scale for women]. J Korean Acad Nurs. 2008 Dec;38(6):813-21. doi: 10.4040/jkan.2008.38.6.813. Korean. PMID 19122483
- [Result] Kim KK, Horan ML, Gendler P, Patel MK. Development and evaluation of the Osteoporosis Health Belief Scale. Res Nurs Health. 1991 Apr;14(2):155-63. doi: 10.1002/nur.4770140210. PMID 2047537
- [Result] Alnuaimi K, Abuidhail J, Abuzaid H. The effects of an educational programme about preeclampsia on women's awareness: a randomised control trial. Int Nurs Rev. 2020 Dec;67(4):501-511. doi: 10.1111/inr.12626. Epub 2020 Sep 22. PMID 32964458
- [Result] Darawad MW, Shawashi TO, Al Duraidi H, Nofal B. Osteoporosis education: Evaluation of an awareness program among female university students. Int J Orthop Trauma Nurs. 2022 May;45:100926. doi: 10.1016/j.ijotn.2022.100926. Epub 2022 Feb 11. PMID 35427994
- [Result] Erenoglu R, Yaman Sozbir S. The Effect of Health Education Given to Syrian Refugee Women in Their Own Language on Awareness of Breast and Cervical Cancer, in Turkey: a Randomized Controlled Trial. J Cancer Educ. 2020 Apr;35(2):241-247. doi: 10.1007/s13187-019-01604-4. PMID 31414370
- [Result] Pınar G, Pınar T. The Impact of health belief model based educational ıntervention on women's knowledge, beliefs, preventive behaviors and clinical outcomes about osteoporosis. SAGE Open. 2020; 10(3), 2158244020941473.
- [Result] Akürk SO, Meseri R, & Özentürk, MG. The psychometric property evaluation of the turkish version of the osteoporosis awareness scale. Turkish Journal of Osteoporosis/Turk Osteoporoz Dergisi. 2021; 27(3), 151-158.
- [Result] ATEŞMAN, E. Türkçe'de okunabilirliğin ölçülmesi. A.Ü. Tömer Dil Dergisi. 1997; 58: 71-74
- [Result] Kılıç D, Erci B. Osteoporoz sağlık inanç ölçeği, osteoporoz öz-etkililik/yeterlik ölçeği ve osteoporoz bilgi testi'nin geçerlilik ve güvenirliği. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi. 2004; 7(2); 89-102.
- [Result] Gökdoğan F."Etkili bir hasta iletişimi için araç geliştirme: yazılı materyallerin uygunluğunun Değerlendirilmesi (DISCERN). Onkoloji Hemşireliği Derneği Bülteni.2003; 16-17: 8-16
- [Result] Oz Yildirim O, Aydin Avci I, Yildirim E, Bostanci Y. The effect of the Incontinence Health Belief Development Program on women's urinary incontinence awareness and health beliefs: a randomized controlled trial. Int Urogynecol J. 2023 Jul;34(7):1385-1393. doi: 10.1007/s00192-022-05343-x. Epub 2022 Sep 21. PMID 36129479